CLINICAL TRIAL: NCT05789771
Title: Abemaciclib Combined With Endocrine Therapy or as a Single Agent for the Treatment of Luminal Metastatic breAst caNcer in the Real-life Clinical pracTice in Russia. Prospective, Multicentre, Non-interventional, Observational Study.
Brief Title: Abemaciclib for the Treatment of Luminal Metastatic breAst caNcer in the Real-life Clinical pracTice in Russia.
Acronym: ATLANT
Status: Completed | Type: Observational
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Collaborators: Russian Society of Clinical Oncology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 15.03.2023
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: HR+/HER2- Breast Cancer; Metastatic Disease; Аdvanced Disease
Keywords: HR+/HER2- breast cancer; abemaciclib
MeSH Terms: conditions — Neoplasm Metastasis | interventions — abemaciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with HR+/HER2- ABC/MBC who received abemaciclib based therapy for their ABC/MBC.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Abemaciclib 150 mg orally every 12 hours plus Aromatase Inhibitor ( Anastrozole 1 mg, Letrozole 2.5 mg or exemestane 25 mg orally every 24 hours on Days 1 to 28 of a 28-day cycle)
  Other Names: VERZENIO
Drug: Abemaciclib — Abemaciclib 150 mg orally every 12 hours plus Fulvestrant (500 mg intramuscularly on Days 1 and 15 of Cycle 1, then on Day 1 of Cycle 2 and beyond on Day 1 of a 28-day cycle)
  Other Names: VERZENIO
Drug: Abemaciclib — Abemaciclib 200 mg orally every 12 hours
  Other Names: VERZENIO

SUMMARY:
The ATLANT study is prospective, multicentre, non-interventional, observational study. Patients with HR+/HER2-negative metastatic breast cancer received abemaciclib as monotherapy or in combination with endocrine therapy.

DETAILED DESCRIPTION:
The ATLANT study is prospective, multicentre, non-interventional, observational study.

136 patients with HR+/HER2-negative metastatic breast cancer received abemaciclib as monotherapy or in combination with endocrine therapy in different line therapy.

The purpose of this study is to better understand how abemciclib combinations are used in real-life conditions and their clinical impact for the treatment of Russian patients affected by (HR+)/ (HER2-) advanced breast cancer (ABC) or metastatic breast cancer (MBC).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients must have a diagnosis of HR+ breast cancer. To fulfill the requirement of HR+ disease, a breast cancer must express, by immunohistochemistry (IHC), at least one of the hormone receptors (ER, progesterone receptor [PgR]) as defined in the relevant American Society of Clinical Oncology/College of American Pathologists Guidelines: For ER and PgR assays to be considered positive, ≥1% of tumor cell nuclei must be immunoreactive by immunohistochemistry (IHC)
3. Patient has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing.
4. Patients with advanced (loco-regionally recurrent, or metastatic) breast cancer not amenable to curative therapy.
5. WHO performance status of 0-2
6. The patient has adequate organ function
7. Any number of prior therapies (including none) is permitted
8. Рatients who will start Abemaciclib as a Single Agent or in combination with endocrine therapy

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, known ongoing or active infection, including HIV, active hepatitis B or C, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (specifically, atrial fibrillation or ventricular dysrhythmias except ventricular premature contractions), or psychiatric illness/social situations that would limit compliance with study requirements.
2. Participants must not be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed HR-positive, HER2-negative breast cancer treated with abemaciclib in combination with endocrine therapy or as a single agent
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) of patients receiving abemaciclib | Up to 5 years
  Progression-free Survival (PFS) of patients receiving abemaciclib in combination with endocrine therapy
  Progression-free Survival (PFS) of patients receiving abemaciclib as a single agent

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 5 years
  ORR is defined as the proportion of patients with best overall response of CR or PR according to RECIST 1.1.
Time To Chemotherapy (TTC) | Up to 5 years
  TTC is defined as the time from date of start of treatment to the date of the first documented chemotherapy
Time To New Treatment Options (TTN) | Up to 5 years
  TTN s defined as the time from date of start of treatment to the date of the first new New Treatment Options
Frequency of AE/SAE | Up to 5 years
  occurenec of AE/SAE during therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Russian Society of Clinical Oncology, Moscow, Russia